CLINICAL TRIAL: NCT05836077
Title: Education Given to Breast Cancer Patients Receiving Chemotherapy With Pecha Kucha Method Effects on Posttraumatic Growth and Psychological Resilience
Brief Title: Pecha Kucha Method Effects on Posttraumatic Growth and Psychological Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/ 03- 24
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Growth; Psychological Resilience; Breast Cancer Patients
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Pecha kucha method and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecha kucha method (Experimental): Patients will be trained by pecha kucha method using computer with powepoint presentation.
  Interventions: Other: Education with pecha kucha method
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Education with pecha kucha method — Education with pecha kucha method
  Arms: Pecha kucha method

SUMMARY:
This study was planned to investigate the effect of the training given to breast cancer patients receiving chemotherapy with pecha kucha method on posttraumatic growth and psychological resilience.

DETAILED DESCRIPTION:
This study is a randomized controlled trial planned to investigate the effect of the training given to breast cancer patients receiving chemotherapy with the pecha kucha method on posttraumatic growth and psychological resilience.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* At least one course of adjuvant chemotherapy prior to treatment,
* Literacy
* Communicable patients
* Patients who agreed to participate in the study

Exclusion Criteria:

* With a psychiatric diagnosis,

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients receiving chemotherapy
Enrollment: 90 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Growth Inventory | Before the training
  The 6-point Likert-type scale consists of 21 items and a 5-factor structure and is scored between 0-5. The total score that can be obtained from the scale varies between 0-105. The sub-dimensions of the scale are relationships with others, new possibilities, personal empowerment, spiritual change and appreciation of life. High scores on the scale indicate that posttraumatic growth is high.
Post Traumatic Growth Inventory | 1 month after the training
  The 6-point Likert-type scale consists of 21 items and a 5-factor structure and is scored between 0-5. The total score that can be obtained from the scale varies between 0-105. The sub-dimensions of the scale are relationships with others, new possibilities, personal empowerment, spiritual change and appreciation of life. High scores on the scale indicate that posttraumatic growth is high.
  Before the training
  1 month after the training
The Brief Resilience Scale | Before the training
  The scale measures the psychological resilience of individuals. It is a 5-point Likert-type, 6-item, self-report measurement tool. High scores on the scale indicate high psychological resilience.
The Brief Resilience Scale | 1 month after the training
  The scale measures the psychological resilience of individuals. It is a 5-point Likert-type, 6-item, self-report measurement tool. High scores on the scale indicate high psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Principal Investigator — Istanbul Sabahattin Zaim University
Locations (1):
- Zülfünaz Özer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakir N, Gun Kakasci C, Demir C. The effect of training with the Pecha Kucha method on the attitudes of chronically ill women toward COVID-19 vaccination. Women Health. 2022 Oct-Dec;62(9-10):809-817. doi: 10.1080/03630242.2022.2146834. Epub 2022 Nov 14. PMID 36377268